CLINICAL TRIAL: NCT07283809
Title: European Unified Registries for Heart Care Evaluation and Randomised Trials
Brief Title: European Unified Registries for Heart Care Evaluation and Randomised Trials Italy
Acronym: EuroHeart ITA
Status: Recruiting | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K27
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: ACS - Acute Coronary Syndrome
Keywords: Quality indicators; ACS; STEMI; NSTEMI; ESC; Guidelines
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adherence to European Society of Cardiology (ESC) quality indicators — EuroHeart is an initiative of the European Society of Cardiology (ESC) supporting continuous quality-of-care improvement through individual patient data collection. The present registry component refers specifically to the Italian implementation of the EuroHeart programme, aimed at monitoring and improving adherence to ESC quality indicators within Italian clinical practice.

SUMMARY:
Major advances in cardiovascular medicine have been driven by innovations in basic research in biological and technical sciences. Despite the clear evidence regarding the treatments that have been demonstrated to be useful to improve patients' outcomes, their transferability to everyday clinical practice seems to be at least suboptimal. The European Society of Cardiology (ESC), therefore, planned to support a program, denominated EuroHeart, for continuous data collection of standardized and/or harmonized variables in common cardiovascular diseases, such as ACS, HF and A Fib. EuroHeart is an observational, prospective, multicentre initiative with continuous data collection in consecutive patients with ACS, HF and A Fib to support continuous quality of care improvement through the evaluation of quality indicators (QIs) defined by the ESC. All patients included in the EuroHeart initiative, will enter a 12 month longitudinal follow-up with the collection of clinical events and clinical status data.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age.
* Males and females at birth.
* At least one of the following clinical conditions:
* Hospitalization for Acute Coronary Syndrome (ACS)
* Heart failure (HF, outpatients, and/or inpatients)
* Atrial fibrillation (A Fib, outpatients and/or inpatients)
* Signed informed consent for the study and for privacy.

Exclusion Criteria:

* patients who do not sign the consent to participate in the project and/or Privacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ACS
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to ESC Quality indicators (STEMI patients reperfused) | From enrollment to 12 months follow-up
  Proportion of patients with STEMI reperfused among those eligible (onset of symptoms to diagnosis <12 hours)
Adherence to ESC Quality indicators (STEMI patients reperfused <90 min) | From enrollment to 12 months follow-up
  Proportion of patients with STEMI who receive timely reperfusion with PCI (wire crossing) within 90 minutes from initial diagnostic ECG
Adherence to ESC Quality indicators (coronary angiography in NSTEMI patients within 24 hours) | From enrollment to 12 months follow-up
  Rate of NSTEMI patients who receive invasive within 24 hours from their diagnosis
Adherence to ESC Quality indicators (radial access) | From enrollment to 12 months follow-up
  Use of radial access in case of invasive strategy for patients with STEMI and NSTEMI
Adherence to ESC Quality indicators (time to reperfusion in STEMI patients) | From enrollment to 12 months follow-up
  The time between the initial STEMI diagnosis and arterial access (absolute value) for primary PCI
Adherence to ESC Quality indicators (pre-discharge LVEF evaluation in STEMI and NSTEMI patients) | From enrollment to 12 months follow-up
  The proportion of patients with STEMI and NSTEMI who have an assessment of their left ventricular ejection fraction (LVEF) before hospital discharge
Adherence to ESC Quality indicators (in hospital LDL-c evaluation in STEMI and NSTEMI patients) | From enrollment to 12 months follow-up
  The proportion of patients with STEMI and NSTEMI who have their LDL cholesterol measured during hospitalization
Adherence to ESC Quality indicators (DAPT prescription at discharge in STEMI and NSTEMI patients) | From enrollment to 12 months follow-up
  Proportion of patients with STEMI and NSTEMI discharged on dual antiplatelet therapy
Adherence to ESC Quality indicators (LLA prescription at discharge in STEMI and NSTEMI patients) | From enrollment to 12 months follow-up
  Proportion of patients discharged from hospital on Lipid Lowering Agents (LLA)
Adherence to ESC Quality indicators (ACEi/ARB/ARNI prescription at discharge in patients with LVEF ≤40%) | From enrollment to 12 months follow-up
  Proportion of patients with LVEF ≤40% who are discharged from hospital on angiotensin converting enzymes inhibitors (ACEi) or angiotensin receptor blockers (ARBs) or angiotensin receptor-neprilysin inhibitor (ARNI)
Adherence to ESC Quality indicators (Beta blockers prescription at discharge in patients with LVEF ≤40%) | From enrollment to 12 months follow-up
  Proportion of patients with LVEF ≤40% who are discharged from hospital on beta blockers.

SECONDARY OUTCOMES:
Cardiovascular and non-cardiovascular events during follow-up | 12 months follow-up
  Proportion of patients with clinical events at 12 months

CONTACTS AND LOCATIONS:
Locations (57):
- Italy (57):
  - Ospedale Valdarno S. Maria Della Gruccia - U.O. Malattie Cardiovascolari, Montevarchi, AREZZO
  - Ospedale Miulli - U.O.C. Cardiologia - Utic, Acquaviva delle Fonti, BA
  - Ospedale Della Murgia - Fabio Perinei - S.C. Cardiologia-Utic, Altamura, BA
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Ospedale Di Venere - U.O.C. Di Cardiologia, Bari, BA
  - Asst Spedali Civili - Cardiologia, Brescia, BS
  - A.O.U. Cagliari Policlinico Monserrato - Sc Cardiologia Utic Emodinamica, Monserrato, CAGLIARI
  - Azienda Ospedaliera Cannizzaro - Uoc Cardiologia, Catania, CATANIA
  - Ospedale A. Cardarelli - U.O. Cardiologia E Utic, Campobasso, CB
  - Azienda Ospedaliera S. Anna E S. Sebastiano - U.O. Cardiologia D'Emergenza Con Utic, Caserta, CE
  - Casa Di Cura San Michele - Uo Cardiologia, Maddaloni, CE
  - Ospedale Di Cremona - Uo Di Cardiologia, Cremona, CR
  - Ospedale Civile Ferrari - U.O.C. Cardiologia-Utic, Castrovillari, CS
  - Ospedale Annunziata - Uoc Cardiologia, Cosenza, CS
  - P.O. "Pugliese" - A.O.U. "Renato Dulbecco" - Utic-Emodinamica E Cardiologia Interventistica, Catanzaro, CZ
  - Policlinico Riuniti - S.C. Di Cardiologia Universitaria-Utic, Foggia, FG
  - Ospedale San Giuseppe - Cardiologia, Empoli, FI
  - Aou Careggi - Interventistica Cardiologica Strutturale, Florence, FI
  - Irccs Ospedale Policlinico San Martino - Unita' Operativa Cardiologia, Genova, GE
  - Irccs Centro Neurolesi Bonino Pulejo - P.O. Piemonte - Cardiologia E Utic, Messina, MESSINA
  - Policlinico G. Martino U.O.C - Cardiologia Con Utic, Messina, MESSINA
  - Ospedale Civile Fornaroli - U.O. Cardiologia, Magenta, MILANO
  - Irccs Ospedale San Raffaele - Area Unica Di Terapia Intensiva Cardiologica E Cch, Milan, MILANO
  - Ospedale L. Sacco - Sc Cardiologia, Milan, MILANO
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 1 - Emodinamica, Milan, Mlano
  - Aou Federico Ii - Uoc Cardiologia Emodinamica Ed Utic, Napoli, NAPOLI
  - Aou Policlinico P. Giaccone - U.O.C. Cardiologia, Palermo, PALERMO
  - Aor Villa Sofia-Cervello Po Villa Sofia - Uoc Cardiologia E Utic E Emodinamica -Villa Sofia, Palermo, PALERMO
  - Azienda Ospedale-Universita Padova - Uosd Terapia Intensiva Cardiologica, Padua, PD
  - Ospedale Civile Dello Spirito Santo - Cardiologia Con Utic, Pescara, PE
  - Azienda Ospedaliera Di Perugia - S.C. Cardiologia, Perugia, PG
  - Ospedale Civile - U.O.C. Cardiologia - Utic, Fidenza, PR
  - Presidio Ospedaliero San Salvatore - Cardiologia E Utic, Pesaro, PU
  - Po Santa Maria Nuova - Ausl Re Irccs - Soc Cardiologia Ospedaliera, Reggio Emilia, RE
  - Ospedale Giovanni Paolo Ii - U.O.C. Cardiologia-Utic, Ragusa, RG
  - P.O. San Camillo de Lellis - U.O.C. Cardiologia, Rieti, RIETI
  - Campus Biomedico - Cardiologia, Roma, RM
  - P.O. San Filippo Neri - Asl Roma 1 - Cardiologia Intensiva Ed Interventistica, Roma, RM
  - Ospedale Sandro Pertini - Uoc Cardiologia - Utic, Roma, RM
  - Policlinico Casilino - U.O.C. Cardiologia, Roma, RM
  - Ospedale Madre Giuseppina Vannini - U.O.C. Cardiologia, Roma, RM
  - Ospedale Santa Maria Della Misericordia - U.O.C. Cardiologia, Rovigo, RO
  - Ospedale San Luca - U.O. Utic - Cardiologia, Vallo della Lucania, SA
  - Aou Senese Ospedale S. Maria Alle Scotte - Cardiologia, Siena, SI
  - P.O. Levante - Ospedale San Paolo - S.C. Cardiologia Levante, Savona, SV
  - Ospedale Civile - S.C. Cardiologia, Ivrea, TO
  - Aou Citta' Della Salute E Della Scienza - S.C. Cardiologia U, Torino, TO
  - Ospedale Santa Maria Del Carmine - U.O. Cardiologia Ad Indirizzo Elettrofisiologia, Rovereto, TRENTO
  - Ospedale Santa Chiara - Divisione Di Cardiologia, Trento, TRENTO
  - Asugi - Ospedale Di Cattinara - S.C. Cardiologia, Trieste, TS
  - Ospedale Ca' Foncello - U.O.C. Cardiologia, Treviso, TV
  - Pou "Santa Maria Della Misericordia" - S.O.C. Cardiologia, Udine, UD
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VARESE
  - Ospedale Civile - U.O.C. Di Cardiologia, Arzignano, VI
  - Irccs Ospedale Sacro Cuore Don Calabria - U.O. Di Cardiologia, Negrar, VR
  - Aoui Di Verona - U.O. Cardiologia, Verona, VR
  - Aou Maggiore Della Carita' - Ssvd Utic, Novara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schiele F, Aktaa S, Rossello X, Ahrens I, Claeys MJ, Collet JP, Fox KAA, Gale CP, Huber K, Iakobishvili Z, Keys A, Lambrinou E, Leonardi S, Lettino M, Masoudi FA, Price S, Quinn T, Swahn E, Thiele H, Timmis A, Tubaro M, Vrints CJM, Walker D, Bueno H; ESC Scientific Document Group; Halvorsen S, Jernberg T, Jortveit J, Blondal M, Ibanez B, Hassager C. 2020 Update of the quality indicators for acute myocardial infarction: a position paper of the Association for Acute Cardiovascular Care: the study group for quality indicators from the ACVC and the NSTE-ACS guideline group. Eur Heart J Acute Cardiovasc Care. 2021 Apr 8;10(2):224-233. doi: 10.1093/ehjacc/zuaa037. PMID 33550362
- [Background] Batra G, Aktaa S, Camm AJ, Costa F, Di Biase L, Duncker D, Fauchier L, Fragakis N, Frost L, Hijazi Z, Juhlin T, Merino JL, Mont L, Nielsen JC, Oldgren J, Polewczyk A, Potpara T, Sacher F, Sommer P, Tilz R, Maggioni AP, Wallentin L, Casadei B, Gale CP. Data standards for atrial fibrillation/flutter and catheter ablation: the European Unified Registries for Heart Care Evaluation and Randomized Trials (EuroHeart). Eur Heart J Qual Care Clin Outcomes. 2023 Sep 12;9(6):609-620. doi: 10.1093/ehjqcco/qcac068. PMID 36243903
- [Background] Aktaa S, Batra G, Cleland JGF, Coats A, Lund LH, McDonagh T, Rosano G, Seferovic P, Vasko P, Wallentin L, Maggioni AP, Casadei B, Gale CP; Heart Failure Association of the European Society of Cardiology. Data standards for heart failure: the European Unified Registries for Heart Care Evaluation and Randomized Trials (EuroHeart). Eur Heart J. 2022 Jun 14;43(23):2185-2195. doi: 10.1093/eurheartj/ehac151. PMID 35443059
- [Background] Association of Cardiovascular Nursing and Allied Professions (ACNAP); Association for Acute CardioVascular Care (ACVC); European Association of Percutaneous Cardiovascular Interventions (EAPCI); EURObservational Research Programme (EORP); ESC Patient Forum; ESC Working Group on Thrombosis and ESC Committee for Young Cardiovascular Professionals; Batra G, Aktaa S, Wallentin L, Maggioni AP, Ludman P, Erlinge D, Casadei B, Gale CP. Data standards for acute coronary syndrome and percutaneous coronary intervention: the European Unified Registries for Heart Care Evaluation and Randomised Trials (EuroHeart). Eur Heart J. 2022 Jun 21;43(24):2269-2285. doi: 10.1093/eurheartj/ehac133. PMID 35380662
- [Background] Aktaa S, Batra G, Wallentin L, Baigent C, Erlinge D, James S, Ludman P, Maggioni AP, Price S, Weston C, Casadei B, Gale CP. European Society of Cardiology methodology for the development of quality indicators for the quantification of cardiovascular care and outcomes. Eur Heart J Qual Care Clin Outcomes. 2022 Jan 5;8(1):4-13. doi: 10.1093/ehjqcco/qcaa069. PMID 32845314
- [Background] Wallentin L, Gale CP, Maggioni A, Bardinet I, Casadei B. EuroHeart: European Unified Registries On Heart Care Evaluation and Randomized Trials. Eur Heart J. 2019 Sep 1;40(33):2745-2749. doi: 10.1093/eurheartj/ehz599. No abstract available. PMID 31505603